CLINICAL TRIAL: NCT00871845
Title: Effects of Dietary and Behavioral Intervention and Orlistat for Management of Obesity and Metabolic Syndrome on Response to Hepatitis C Therapy
Brief Title: Increasing Cure Rate of Hepatitis C Therapy in Obese Hepatitis C Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol expired and not renewed
Sponsor: Hossam Kandil (Other)
Responsible Party: Sponsor-Investigator, Hossam Kandil, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO07090035
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Insulin Resistance; Metabolic Syndrome; Hepatitis C
Keywords: obesity; hepatitis C; insulin resistance; metabolic syndrome
MeSH Terms: conditions — Obesity; Insulin Resistance; Metabolic Syndrome; Hepatitis C | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Both groups followed for same period of time
Masking Description: Participants were divided into arms based upon BMI. Weight loss instruction/management provided only to overweight arm.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LEAN (non obese, naive) (No Intervention): Patients naive to hepatitis C therapy with body mass index (BMI) <25
- OVERWEIGHT (obese, naive, control) (Other): Patients naive to hepatitis C therapy with BMI ≥ 25, received Dietary and Lifestyle modification educational sessions (one-time 15 minute weight loss instruction and pamphlet and enrolled into weight management program with 5 weekly one-hour nutrition and physical exercise education sessions after initial evaluation followed by monthly follow up.)
  Interventions: Behavioral: Dietary and Lifestyle modification educational sessions

INTERVENTIONS:
Behavioral: Dietary and Lifestyle modification educational sessions — 6 sessions of dietary and physical education after which they will start receiving their standard hepatitis C treatment. they will be encouraged to attend up to 12 monthly meetings (along side the monthly visits for their standard viral hepatitis therapy.
  Other Names: weight management classes; weight reduction counseling
  Arms: OVERWEIGHT (obese, naive, control)

SUMMARY:
The purpose of this study is to determine whether obese people do not respond to hepatitis C treatment as well as lean people. This research studies whether obese people will show higher sustained virologic response rate if they lose weight by Orlistat use and dietary and lifestyle modification.

DETAILED DESCRIPTION:
This study is designed to be an interventional, prospective, randomized, double-blinded case-control clinical trial. Procedures will be done in the Center for Liver Diseases, 9'Th floor of Kaufmann medical building, UPMC, USA. This study will also be carried out in National Liver Institute, Egypt.

For treatment-naïve patients, we are targeting 32 subjects for each group; however, we are going to include 37 in each group to allow for estimated drop-outs rate of 15%. Subjects will be randomly assigned to 4 groups as follows: Group 1 includes non-obese controls (BMI < 25). They will receive one session of dietary and behavioral education. Groups 2, 3 and 4 include obese subjects (BMI ≥ 30). Group 2 includes obese controls who will receive one session of dietary and behavioral education. Groups 3 and 4 will receive up to 6 weekly sessions followed by 12 monthly sessions of dietary and behavioral education. Orlistat and placebo will be prescribed for Groups 3 and 4 respectively.

For non-responders and releasers to previous anti-hepatitis C therapy who have BMI ≥ 25 (overweight or obese), subjects will be randomized to groups 5 and 6 and will receive same treatment as groups 3 and 4, respectively. Their results will be compared to the historic controls results.

Screening procedures:

Verifying the eligibility of patients for participation in the study will be done through reviewing data in medical history, physical examination and investigations included in the patients' medical records. Acquired immuno-deficiency syndrome (AIDS) status of the participating subject will be determined by reviewing HIV ELISA screening test, reported in the subject's medical records as well. Measurements of weight and height (for BMI calculation) will be taken and recorded during the initial clinic visit at the center for liver diseases for all patients who agree to participate and fulfill the inclusion and exclusion criteria. Weight measure will be taken while patient is in light underwear and without shoes, while standing with his arms lying alongside the body, and in apnea fixed at midexpiratory phase while height measure will be taken by a wall-mounted stadiometer and recorded to the nearest cm.

Experimental procedures:

Subjects will be randomly grouped into groups by simple randomization method. One of the investigators will pick one folded paper out of a plastic bag that contains folded papers labeled on the folded side with the number of the group.

Further randomization will be done in the pharmacy by the same way to include treatment naïve candidates to groups 3 and 4 and to include treatment non naïve candidates to groups 5 and 6. Therefore, study team will be blinded from type of drug which the candidate will receive, whether Orlistat or placebo, respectively.

Groups 1 and 2 as control groups will receive one session of dietary and physical education, and then they will start receiving standard hepatitis C treatment.

Groups 3, 4, 5 and 6 as interventional groups will receive up to 6 sessions of dietary and physical education after which they will start receiving their standard hepatitis C treatment. Groups 3 and 4 will be encouraged to attend up to 12 monthly meetings (along side the monthly visits for their standard viral hepatitis therapy) at the health education room of center for liver diseases, to check dietary diaries and patient records of physical activity, discuss any related issues, reinforce and encourage compliance to dietary and physical exercise recommendations. The dietary and physical education (given through up to 6 weekly sessions and subsequently up to 12 monthly follow-up meetings) will be presented. It will be based on previously reported (Kelley et al. 2004) lifestyle modifications and dietary regulation program that includes healthy food selections, emphasizing reduced fat consumption (<=30% of daily calories) and restriction of portions to create a daily negative energy balance of ~500 kcal/day. Participants will be encouraged to start with 10 minutes of physical activity such as walking or cycling then gradually increase the activity duration up to 30 minutes. The dietitian will provide each subject with diary for daily recording of dietary intake.

Orlistat (60 mg capsules, three times daily, before meals)will be prescribed for groups 3 and 5. Placebo will be administered for groups 4 and 6. Orlistat or Placebo will be given for 3 to 6 weeks prior to and during the 48 weeks of the standard anti-viral therapy. Pill counts will be obtained monthly to monitor medication compliance.

Stress assessment will be done for the study candidates through a stress specific questionnaire before the start of the study and every 12 weeks afterwards.

Stool samples will be taken from all patients before they start Interferon therapy and every 12 weeks on therapy. Stool samples will be stored at -80 degree Celsius for future PCR study of fecal micro flora.

Follow-up procedures:

Virological and biochemical responses will be followed as clinically indicated by clinical provider. Anthropometric measures of obesity such as measurements of weight, height (for BMI calculation), waist circumference, hip circumference, skin fold thickness and mid-arm circumference will be monthly followed and recorded. Midarm circumference and triceps skin fold thickness will be measured on the left arm midway between the tip of the acromion and the tip of olecranon and was recorded to the nearest 5 cm. Skin fold thickness will be measured at triceps. Waist circumference will be measured midway between iliac crest and lowest rib margin, and hip circumference at the level of the greater trochanters (Han et al. 2001).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* positive diagnosis of hepatitis C, by Polymerase Chain Reaction (PCR
* scheduled to start treatment of hepatitis C by peg interferon and ribavirin
* agreeing to give a written consent to participate in this study.

Exclusion Criteria:

* patients under 18 years of age
* refusal to give a consent to participate in the study
* history of recreational drug or alcohol use in the preceding 6 months
* pregnancy by hCG pregnancy testing which will be done prior to and monthly during the 12 month hepatitis C therapy and for 6 months following the end of treatment
* plan for pregnancy during the study period
* failure to adhere to contraceptive methods
* HIV disease
* evidence of cirrhosis or confirmed hepatocellular carcinoma (HCC), evidence of decompensated liver disease or presence of other liver diseases such as hepatitis B, hemochromatosis, autoimmune hepatitis and Wilson disease
* Patients will be removed from the study if they develop severe side effects to IFN (e.g marked depression, autoimmune reactions like thyroiditis, aplastic anemia..), severe side effects to ribavirin (e.g. marked hemolysis) or intolerance of Orlistat/placebo (e.g. allergic reaction, diarrhea, flatulence..) and withdrawal of the consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hossam M Kandil, MD, PhD, Principal Investigator — assistant professor of medicine
Locations (1):
- Center for Liver Diseases, UPMC., Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While the initial study design included a drug intervention, drug intervention was not done. The study team could not identify an adequate study population willing to undergo drug intervention and funding to cover the costs of the drug intervention. Therefore, the only intervention was weight loss instruction/management.
Groups:
- Lean: Treatment naive HCV Genotype 1 infected patients with BMI<25
- Overweight: Treatment naive HCV Genotype 1 infected patients with BMI >=25
Period: Overall Study
Arm/Group | Lean | Overweight
Started | 11 | 25
Completed | 11 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lean: Lean (BMI<25)
- Overweight: Overweight (BMI>=25)
- Total: Total of all reporting groups
Arm/Group | Lean | Overweight | Total
Number analyzed (Participants) | 11 | 25 | 36
Age, Customized [Count of Participants; unit: Participants]
  Age > 50 years | 4 | 20 | 24
  Age ≤ 50 years | 7 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 4 | 11 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HCV RNA (Early Virological Response)
Description: Early virological response (EVR) defined as a greater than 2-log10 decline in serum HCV RNA from the pretreatment baseline or an undetectable serum HCV RNA at treatment week 12
Time Frame: Week 12
Measure: Number; unit: percentage of participants
Arm/Group | Lean | Overweight
Number analyzed (Participants) | 11 | 25
percentage of participants | 82 | 52

2. Primary Outcome: Body Weight Loss
Description: Mean weight change from week 0 to week 12
Time Frame: Weight loss as of Week 12
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Lean: Lean (BMI < 25)
- Overweight: Overweight (BMI >=25)
Arm/Group | Lean | Overweight
Number analyzed (Participants) | 11 | 25
kg | 1.44 (3.82) | 3.44 (4.12)

3. Primary Outcome: Percentage of Participants With Early Virological Response (EVR) and Significant Weight Loss
Description: EVR compared between overweight subjects who achieved significant weight loss (>=3%) and those who did not
Time Frame: Week 12
Measure: Number; unit: percentage of participants
Groups:
- Overweight Achieving >= 3% Weight Loss: Overweight subjects who achieved significant weight loss (>=3%)
- Overweight Not Achieving >=3% Weight Loss: Overweight subjects who did NOT achieve significant weight loss (>=3%)
Arm/Group | Overweight Achieving >= 3% Weight Loss | Overweight Not Achieving >=3% Weight Loss
Number analyzed (Participants) | 15 | 10
percentage of participants | 69 | 33

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Collected AEs related to nutrition and exercise interventions, not Hepatitis C therapy
Arm/Group | Lean | Overweight
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/25
Other Adverse Events (participants affected / at risk) | 0/11 | 0/25

LIMITATIONS AND CAVEATS:
Study design adjusted due to subject availability & financial constraints. The drug intervention was not done. Waist circum & skin fold thickness not done due to patient refusal. HOMA/IR not done as not available/performed by primary providers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No